CLINICAL TRIAL: NCT04075461
Title: Is arthroplaSty bEtter Than interNal Fixation in the undiSplaced Femoral nEck Fracture? A National Pragmatical Randomized Controlled Trial - the SENSE Trial
Brief Title: Arthroplasty Versus Internal Fixation for Undisplaced Femoral Neck Fracture
Acronym: SENSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Aalborg University Hospital (Other); Regionshospital Nordjylland (Other Government); Aarhus University Hospital (Other); Odense University Hospital (Other); Slagelse Hospital (Other); Bispebjerg Hospital (Other); Regionshospitalet Viborg, Skive (Other); Randers Regional Hospital (Other); Regionshospitalet Horsens (Other); Hospital of Southern Jutland (Other); Esbjerg Hospital - University Hospital of Southern Denmark (Other); Hvidovre University Hospital (Other); Herlev Hospital (Other); Hillerod Hospital, Denmark (Other); Holbaek Sygehus (Other); Zealand University Hospital (Other); Sygehus Lillebaelt (Other); Nykøbing Falster County Hospital (Other); Regional Hospital West Jutland (Other); Bornholm Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S-20180036
Record Dates: First submitted 2019-08-22; First posted 2019-08-30 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Undisplaced Fracture; Femoral Neck Fractures; Internal Fixation; Complications; Arthroplasty Complications
MeSH Terms: conditions — Femoral Neck Fractures | interventions — Arthroplasty; Fracture Fixation, Internal

STUDY DESIGN:
Intervention Model Description: The study is designed as a national pragmatical RCT including all patients with an undisplaced FNF and a NMS score of 5 and above. The standard treatment in Denmark is internal fixation and the patients are randomized to arthroplasty or IF. The steering group have assessed the pragmatic attitude of the design and the study reaches 5 points in 7 of the 9 domains (Figure 1) (9). Reporting is performed accordingly to the extension of the CONSORT statements for pragmatical RCT (17). Using the PRECIS-2 we scored the study to 43 points out of 45 possible.
Who Masked: Outcomes Assessor
Masking Description: The surgeon, theater staff and patient cannot be blinded due to the nature of two very different types of surgery. However, the assessors will be blinded for type of surgery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Undisplaced FNF + Arthroplasty (Experimental): Arthroplasty is the typical surgery for a displaced femoral neck fracture
  Interventions: Procedure: Arthroplasty
- Undisplaced FNF + Internal fixation (Active Comparator): Internal fixation is the typical surgery for an undisplaced femoral neck fracture
  Interventions: Procedure: Internal fixation

INTERVENTIONS:
Procedure: Arthroplasty — Arthroplasty is commonly used for a displaced femoral neck fracture.
  Arms: Undisplaced FNF + Arthroplasty
Procedure: Internal fixation — Internal fixation is commonly used for undisplaced femoral neck fracture
  Arms: Undisplaced FNF + Internal fixation

SUMMARY:
This is the world's first national orthopedic randomized controlled trial (RCT) involving 19 out of 21 departments in Denmark. Each year, 7,000 patients suffer a hip fracture. This is a severe condition leading to 25% mortality after 1 year and 40% do not recover to the same functional level. The aim is to compare two surgical treatment methods (metal fixation versus artificial hip) in patients above 65 years with an undisplaced femoral neck fracture. The hypothesis is that even though an artificial hip is a larger surgical procedure than metal fixation of the broken bone, the artificial hip is more stable with less pain due the lack of a healing broken bone and therefore leads to a better and quicker mobilization after surgery. Better mobilization is one of the most important factors for decreasing mortality. We have chosen a pragmatic RCT design by using the local departmental implants. We hope that the knowledge from this study will therefore easily be implemented afterwards.

DETAILED DESCRIPTION:
This is the world's first national orthopedic randomized controlled trial (RCT) involving 20 out of 21 departments in Denmark. The aim is to compare two surgical treatment methods (internal fixation (IF) versus arthroplasty) in patients above 65 years with an undisplaced femoral neck fracture (FNF).

Each year, 7,000 patients suffer a hip fracture. This is a severe condition leading to 25% mortality after 1 year and 40% do not recover to the same functional level. Undisplaced FNF is treated with internal fixation in order to aid in fracture healing. However, approximately 10% in Denmark will suffer a reoperation and two RCT's have demonstrated 20-21% reoperations. In comparison, the reoperation frequency was 5-7% for arthroplasty that also demonstrated slightly faster mobilization which is one of the most important factors for decreasing mortality. The hypothesis is therefore that even though arthroplasty is a larger surgery they benefit from the lack of fracture healing, less pain and faster mobilization.

Patients are included in the emergency department and are electronically randomized to either IF or arthroplasty before the surgery. The design is a pragmatic RCT using the implants which are available in the departments. Furthermore, the postoperative treatment protocol is "business as usual" thereby investigating the precise effect of the intervention in real clinical conditions. In addition to a great external validity this allows for easy implemented after study results. The primary outcome is a validated functional score 1 year after surgery and the sample size is calculated to 330 patients. Secondary outcome measures are additional functional assessments and questionnaires, health related quality of life and pain assessment.

We have set up a steering committee consisting of researchers and senior surgeons with a representative from each region. In addition, all but 1 hospital has a representative in project group. The project is therefore anchored in the entire Denmark.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years old
* Undisplaced femoral neck fracture
* Posterior tilt (18) less than 20 degrees
* NMS (13) = 5 and above, indicating an ability to walk
* Cognitive intact in order to achieve informed consent

Exclusion Criteria:

* The fracture is pathological
* The patient does not speak Danish

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 330 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2024-01-26 (Actual); Study Completion 2025-01-26 (Actual)

PRIMARY OUTCOMES:
New Mobility Score (NMS) | 12 months
  NMS score the level of function with a score from 0-9 points. The best score is 9 points.

SECONDARY OUTCOMES:
EuroQol 5 domain 5 level (EQ-5D-5L) | Admission, 3 months, 6 months and 12 months.
  Health related quality of life assessment with a score from 0-1 point. The best score is 1 point
Oxford Hip Score (OHS) | Admission, 3 months, 6 months and 12 months.
  Specific hip function questionnaire with a score from 0-48 points. The best score is 48 points.
Reoperation | Within 1 year after surgery
  New surgery in relation to the primary surgery
Mortality | Within 1 year after surgery
  Mortality
New Mobility Score (NMS) | Admission, 3 and 6 months
  NMS score the level of function with a score from 0-9 points. The best score is 9 points.
Pain Verbal Rating Scale (VRS) | Admission, 2 and 6 weeks, 3, 6, and 12 months
  Patient reported outcome of pain assessment

OTHER OUTCOMES:
New Mobility Score (NMS) | 2 and 5 years
  NMS score the level of function with a score from 0-9 points. The best score is 9 points.
EuroQol 5 domain 5 level (EQ-5D-5L) | 2 and 5 years
  Health related quality of life assessment with a score from 0-1 point. The best score is 1
Reoperation | 2 and 5 years
  New surgery in relation to the primary surgery, given in numbers and percentage
Mortality | 2 and 5 years
  Mortality given in number of deaths and percentage
Pain Verbal Rating Scale (VRS) | 2 and 5 years
  Patient reported outcome of pain assessment of pain from 1 to 10
Oxford Hip Score (OHS) | 2 and 5 years
  Specific hip function questionnaire with a score from 0-48 points. The best score is 48 points.
de Morton Mobility Index (DEMMI) | Admission, 3 months, 6 months, 12 months, 2 and 5 years
  Mobility index with a score from 0-100 points. The best score is 100 points
Barthel-20 | Admission, 3 months, 6 months, 12 months, 2 and 5 years
  Index for activities of daily living with a score from 0-20 points. The best score is 20 points.
Cumulated Cumulated Ambulation Score (CAS) | Admission, 6 and 12 weeks
  Basic mobility score with a score from 0-6 points. The best score is 6 points.
X-ray measurement 1 | First postoperative x-ray during admission and 1 year
  Quality of implant positioning (IMPO) score with a score from 0-6 point. The best score is 6 points

CONTACTS AND LOCATIONS:
Overall Officials: Bjarke Viberg, MD, PhD, Principal Investigator — Department of Orthopaedic Surgery and Traumatology, Lillebaelt Hospital; Ole Brink, MD, PhD, Study Chair — Department of Orthopaedic Surgery and Traumatology, Aarhus University Hospital; Søren Kold, Professor, Study Chair — Department of Orthopaedic Surgery and Traumatology, Aalborg University Hospital; Morten S Larsen, MD, Study Chair — Odense University Hospital; Kristoffer B Hare, MD, PhD, Study Chair — Department of Orthopaedic Surgery and Traumatology, Slagelse Hospital; Henrik Palm, MD, DmSc, Study Chair — Department of Orthopaedic Surgery and Traumatology, Bispebjerg Hospital
Locations (19):
- Denmark (19):
  - Hospital of Southern Jutland, Aabenraa
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus
  - Bispebjerg Hospital, Copenhagen
  - Herlev Hospital, Copenhagen
  - Hvidovre Hospital, Copenhagen
  - Regional Hospital West Jutland, Gødstrup
  - Hospital of North Zealand, Hillerød
  - North Denmark Regional Hospital, Hjørring
  - Holbæk Hospital, Holbæk
  - Randers Regional Hospital, Horsens
  - Lillebaelt Hospital, Kolding
  - Zealand University Hospital, Køge
  - Nykøbing Falster Hospital, Nykøbing Falster
  - Odense University Hospital, Odense
  - Randers Regional Hospital, Randers
  - Bornholm Hospital, Rønne
  - Slagelse Hospital, Slagelse
  - Viborg Regional Hospital, Viborg

IPD SHARING:
Plan to Share IPD: No
Due to Danish regulation direct data sharing is not possible.

REFERENCES:
- [Background] National Institute for Health and Care Excellence. Hip fracture: mangement. Clinical guideline [CG124]. National Institute for Health and Care Excellence; 2011, updated 2017.
- [Background] Roberts KC, Brox WT, Jevsevar DS, Sevarino K. Management of hip fractures in the elderly. J Am Acad Orthop Surg. 2015 Feb;23(2):131-7. doi: 10.5435/JAAOS-D-14-00432. PMID 25624365
- [Background] Lu Q, Tang G, Zhao X, Guo S, Cai B, Li Q. Hemiarthroplasty versus internal fixation in super-aged patients with undisplaced femoral neck fractures: a 5-year follow-up of randomized controlled trial. Arch Orthop Trauma Surg. 2017 Jan;137(1):27-35. doi: 10.1007/s00402-016-2591-9. Epub 2016 Nov 11. PMID 27837321
- [Background] Dolatowski FC, Frihagen F, Bartels S, Opland V, Saltyte Benth J, Talsnes O, Hoelsbrekken SE, Utvag SE. Screw Fixation Versus Hemiarthroplasty for Nondisplaced Femoral Neck Fractures in Elderly Patients: A Multicenter Randomized Controlled Trial. J Bone Joint Surg Am. 2019 Jan 16;101(2):136-144. doi: 10.2106/JBJS.18.00316. PMID 30653043
- [Background] Wamper KE, Sierevelt IN, Poolman RW, Bhandari M, Haverkamp D. The Harris hip score: Do ceiling effects limit its usefulness in orthopedics? Acta Orthop. 2010 Dec;81(6):703-7. doi: 10.3109/17453674.2010.537808. PMID 21110703
- [Background] Gjertsen JE, Fevang JM, Matre K, Vinje T, Engesaeter LB. Clinical outcome after undisplaced femoral neck fractures. Acta Orthop. 2011 Jun;82(3):268-74. doi: 10.3109/17453674.2011.588857. PMID 21619501
- [Background] Zlowodzki M, Brink O, Switzer J, Wingerter S, Woodall J Jr, Petrisor BA, Kregor PJ, Bruinsma DR, Bhandari M. The effect of shortening and varus collapse of the femoral neck on function after fixation of intracapsular fracture of the hip: a multi-centre cohort study. J Bone Joint Surg Br. 2008 Nov;90(11):1487-94. doi: 10.1302/0301-620X.90B11.20582. PMID 18978271
- [Background] Sikand M, Wenn R, Moran CG. Mortality following surgery for undisplaced intracapsular hip fractures. Injury. 2004 Oct;35(10):1015-9. doi: 10.1016/j.injury.2004.01.004. PMID 15351669
- [Background] Loudon K, Treweek S, Sullivan F, Donnan P, Thorpe KE, Zwarenstein M. The PRECIS-2 tool: designing trials that are fit for purpose. BMJ. 2015 May 8;350:h2147. doi: 10.1136/bmj.h2147. No abstract available. PMID 25956159
- [Background] Kristensen PK, Thillemann TM, Soballe K, Johnsen SP. Are process performance measures associated with clinical outcomes among patients with hip fractures? A population-based cohort study. Int J Qual Health Care. 2016 Dec 1;28(6):698-708. doi: 10.1093/intqhc/mzw093. PMID 27591269
- [Background] de Morton NA, Harding KE, Taylor NF, Harrison G. Validity of the de Morton Mobility Index (DEMMI) for measuring the mobility of patients with hip fracture during rehabilitation. Disabil Rehabil. 2013 Feb;35(4):325-33. doi: 10.3109/09638288.2012.705220. Epub 2012 Aug 16. PMID 22897700
- [Background] de Morton NA, Berlowitz DJ, Keating JL. A systematic review of mobility instruments and their measurement properties for older acute medical patients. Health Qual Life Outcomes. 2008 Jun 5;6:44. doi: 10.1186/1477-7525-6-44. PMID 18533045
- [Background] Parker MJ, Palmer CR. A new mobility score for predicting mortality after hip fracture. J Bone Joint Surg Br. 1993 Sep;75(5):797-8. doi: 10.1302/0301-620X.75B5.8376443.
- [Background] Kristensen MT, Foss NB, Kehlet H. [Timed Up and Go and New Mobility Score as predictors of function six months after hip fracture]. Ugeskr Laeger. 2005 Aug 29;167(35):3297-300. Danish. PMID 16138973
- [Background] Kristensen MT, Bandholm T, Foss NB, Ekdahl C, Kehlet H. High inter-tester reliability of the new mobility score in patients with hip fracture. J Rehabil Med. 2008 Jul;40(7):589-91. doi: 10.2340/16501977-0217. PMID 18758678
- [Background] Pedersen TJ, Lauritsen JM. Routine functional assessment for hip fracture patients. Acta Orthop. 2016 Aug;87(4):374-9. doi: 10.1080/17453674.2016.1197534. Epub 2016 Jun 22. PMID 27329799
- [Background] Zwarenstein M, Treweek S, Gagnier JJ, Altman DG, Tunis S, Haynes B, Oxman AD, Moher D; CONSORT group; Pragmatic Trials in Healthcare (Practihc) group. Improving the reporting of pragmatic trials: an extension of the CONSORT statement. BMJ. 2008 Nov 11;337:a2390. doi: 10.1136/bmj.a2390. PMID 19001484
- [Background] Palm H, Gosvig K, Krasheninnikoff M, Jacobsen S, Gebuhr P. A new measurement for posterior tilt predicts reoperation in undisplaced femoral neck fractures: 113 consecutive patients treated by internal fixation and followed for 1 year. Acta Orthop. 2009 Jun;80(3):303-7. doi: 10.3109/17453670902967281. PMID 19634021
- [Background] Schmidt M, Pedersen L, Sorensen HT. The Danish Civil Registration System as a tool in epidemiology. Eur J Epidemiol. 2014 Aug;29(8):541-9. doi: 10.1007/s10654-014-9930-3. Epub 2014 Jun 26. PMID 24965263
- [Background] Kristensen MT. Hip fractures - Functional assessments and factors influencing in-hospital outcome, a physiotherapeutic perspective. Faculty of Medicine: Lund University; 2010.
- [Background] Steihaug OM, Gjesdal CG, Bogen B, Kristoffersen MH, Lien G, Hufthammer KO, Ranhoff AH. Does sarcopenia predict change in mobility after hip fracture? a multicenter observational study with one-year follow-up. BMC Geriatr. 2018 Mar 5;18(1):65. doi: 10.1186/s12877-018-0755-x. PMID 29506481
- [Background] The Danish Interdisciplinary Registry for Hip Fracture. National Annual Report for 2017. The Danish Healthcare Service; 2017 15.05.2017.
- [Derived] Viberg B, Kold S, Brink O, Larsen MS, Hare KB, Palm H; SENSE collaborators. Is arthroplaSty bEtter than interNal fixation for undiSplaced femoral nEck fracture? A national pragmatic RCT: the SENSE trial. BMJ Open. 2020 Oct 10;10(10):e038442. doi: 10.1136/bmjopen-2020-038442. PMID 33040011

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-12-20): https://cdn.clinicaltrials.gov/large-docs/61/NCT04075461/SAP_000.pdf